CLINICAL TRIAL: NCT03404206
Title: A Randomized, Double-Blind, Placebo-Controlled Trial to Compare the Duration of Analgesic Efficacy and Safety of Naproxen Sodium Tablets and Ibuprofen Tablets in Postsurgical Dental Pain
Brief Title: A Trial to Compare the Duration of Analgesic Efficacy and Safety of Naproxen Sodium Tablets and Ibuprofen Tablets in Postsurgical Dental Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 19762; 2017-005049-67 (EudraCT Number)
Record Dates: First submitted 2018-01-12; First posted 2018-01-19 (Actual); Results first posted 2019-07-18 (Actual); Last update posted 2019-07-18 (Actual); Status verified 2019-06

CONDITIONS: Pain, Postoperative
Keywords: Postsurgical pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Naproxen; Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Naproxen Sodium (Aleve, BAY117031) (Experimental): Participants received one single dose of 440 mg naproxen sodium tablets (200 mg x 2 tablets, oral) after randomization
  Interventions: Drug: Naproxen Sodium (Aleve, BAY117031)
- Ibuprofen (Advil) (Active Comparator): Participants received one single dose of 400 mg ibuprofen tablets (200 mg x 2 tablets, oral) after randomization
  Interventions: Drug: Ibuprofen (Advil)
- Placebo (Placebo Comparator): Participants received one single dose of matching placebo tablets (2 tablets, oral) after randomization
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Naproxen Sodium (Aleve, BAY117031) — 220 mg x 2 tablets, oral, single dose
  Arms: Naproxen Sodium (Aleve, BAY117031)
Drug: Ibuprofen (Advil) — 200 mg x 2 tablets, oral, single dose
  Arms: Ibuprofen (Advil)
Drug: Placebo — Matching placebo, 2 tablets, oral, single dose
  Arms: Placebo

SUMMARY:
To compare the duration of analgesic efficacy as determined by the time to rescue medication of a single oral dose of naproxen sodium 440 mg (2 x 220 mg tablets) relative to ibuprofen 400 mg (2 x 200 mg tablets) and placebo over 24 hours in subjects experiencing moderate to severe post-impaction surgery dental pain.

To compare the overall analgesic effect (SPID 0-24) of a single dose of naproxen sodium 440 mg (2 x 220 mg tablets) relative to ibuprofen 400 mg (2 x 200 mg tablets) and placebo.

To compare the overall relief from pain (TOTPAR 0-24) of a single dose of naproxen sodium 440 mg (2 x 220 mg tablets) relative to ibuprofen 400 mg (2 x 200 mg tablets) and placebo.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, ambulatory, male or female volunteers 16-40 years of age;
* Body mass index 18.0 to 30.0 kg/m^2 inclusive;
* Scheduled to undergo surgical removal of at least 2 mandibular partial or full bony impacted third molars. Up to two maxillary third molars may be removed regardless of impaction level. Supernumerary teeth present may also be removed at the discretion of the oral surgeon;
* Mandibular molars must demonstrate modified Demirjian root classification stage D, E, F, G or H;

Exclusion Criteria:

* History of hypersensitivity to naproxen sodium, ibuprofen, nonsteroidal anti-inflammatory drugs (NSAIDS), aspirin, similar pharmacological agents, local anesthetics, rescue medication or components of the investigational products;
* Evidence or history of clinically significant (in the judgment of the investigator) hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic diseases, or malignancies within the last 5 years;
* Relevant concomitant disease such as asthma (exercise induced asthma is permitted)

Ages: 16 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 387 (Actual)
Dates: Start 2018-02-12 (Actual); Primary Completion 2018-07-06 (Actual); Study Completion 2018-07-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Jean Brown Research, Salt Lake City, Utah, United States

REFERENCES:
- [Derived] Cooper SA, Desjardins P, Brain P, Paredes-Diaz A, Troullos E, Centofanti R, An B. Longer analgesic effect with naproxen sodium than ibuprofen in post-surgical dental pain: a randomized, double-blind, placebo-controlled, single-dose trial. Curr Med Res Opin. 2019 Dec;35(12):2149-2158. doi: 10.1080/03007995.2019.1655257. Epub 2019 Aug 27. PMID 31402718
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe — http://www.clinicaltrialsregister.eu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at one center in the United States, between 12 February 2018 (first patient first visit) and 10 July 2018 (last patient last visit).
Pre-assignment Details: Overall, 387 participants completed surgical teeth extraction, and all of them were randomized and received the treatment.
Period: Overall Study
Arm/Group | Naproxen Sodium (Aleve, BAY117031) | Ibuprofen (Advil) | Placebo
Started | 166 | 166 | 55
Completed | 162 | 164 | 55
Not Completed | 4 | 2 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0
Not completed — Lost to Follow-up | 3 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety Population (included all subjects who were randomized and took at least one dose of investigational product)
Groups:
- Total: Total of all reporting groups
Arm/Group | Naproxen Sodium (Aleve, BAY117031) | Ibuprofen (Advil) | Placebo | Total
Number analyzed (Participants) | 166 | 166 | 55 | 387
Age, Continuous [Mean (Standard Deviation); unit: years] | 19.0 (2.96) | 19.0 (2.62) | 19.0 (2.91) | 19.0 (2.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 77 | 89 | 30 | 196
  Male | 89 | 77 | 25 | 191
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 23 | 25 | 10 | 58
  Not Hispanic or Latino | 143 | 141 | 45 | 329
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 148 | 148 | 48 | 344
  Black or African American | 2 | 4 | 1 | 7
  American Indian or Alaska Native | 3 | 4 | 2 | 9
  Asian | 1 | 2 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 1 | 3 | 1 | 5
  Other | 11 | 5 | 2 | 18
Pain Intensity Score [Count of Participants; unit: Participants] — Categorical pain intensity scale - no pain (0), mild pain (1), moderate pain (2), or severe pain (3) was used for pain intensity assessments.
  Participants
    No Pain (0) | 0 | 0 | 0 | 0
    Mild Pain (1) | 0 | 0 | 0 | 0
    Moderate Pain (2) | 69 | 67 | 23 | 159
    Severe Pain (3) | 97 | 99 | 32 | 228

OUTCOME MEASURES:

1. Primary Outcome: Time to First Use of Rescue Medication
Description: Time to first use of rescue medication was estimated using Kaplan-Meier method. If a subject did not take the rescue medication during the treatment period, (s)he was censored at the time of last assessment.
Time Frame: Up to 24 hours
Population: Per-protocol population
Measure: Number; unit: hours
Arm/Group | Naproxen Sodium (Aleve, BAY117031) | Ibuprofen (Advil) | Placebo
Number analyzed (Participants) | 166 | 165 | 54
hours
  Minimum | 1.22 | 1.22 | 1.18
  25th Percentile | 11.017 | 8.267 | 2.117
  50th Percentile | NA — Not estimable due to censored data | 10.533 | 2.533
  75th Percentile | NA — Not estimable due to censored data | 14.117 | 12.100
  Maximum | 22.17 | 18.28 | 21.75
Statistical Analysis 1: Comparison: Naproxen Sodium (Aleve, BAY117031) vs Ibuprofen (Advil); Test type: Superiority; p < 0.001, Log Rank
Statistical Analysis 2: Comparison: Naproxen Sodium (Aleve, BAY117031) vs Placebo; Test type: Superiority; p < 0.001, Log Rank

2. Secondary Outcome: Sum of Pain Intensity Difference (SPID)
Description: Pain intensity was measured using Numerical Rating Scale (from 0 to 10: 0 = no pain, 10 = worst possible pain). For each postdose time point, pain intensity differences (PIDs) were derived by subtracting the pain intensity at the postdose time point from the baseline intensity score (baseline score - post-baseline score). A positive difference was indicative of improvement. Time-weighted sum of pain intensity differences (SPIDs) were calculated by multiplying the PID score at each postdose time point by the duration (in hours) since the preceding time point and then summing these values.
Time Frame: Up to 24 hours
Population: Per-protocol population
Measure: Mean (Standard Deviation); unit: Scores on a scale * hours
Arm/Group | Naproxen Sodium (Aleve, BAY117031) | Ibuprofen (Advil) | Placebo
Number analyzed (Participants) | 166 | 165 | 54
Scores on a scale * hours | 83.29 (57.177) | 48.54 (40.705) | 9.96 (58.197)
Statistical Analysis 1: Comparison: Naproxen Sodium (Aleve, BAY117031) vs Ibuprofen (Advil); Test type: Superiority; ANCOVA; Least squares means = -34.73, 95% CI 2-sided [-45.67 to -23.8]
Statistical Analysis 2: Comparison: Naproxen Sodium (Aleve, BAY117031) vs Placebo; Test type: Superiority; ANCOVA; Least squares means = -73.43, 95% CI 2-sided [-89.01 to -57.85]
Statistical Analysis 3: Comparison: Ibuprofen (Advil) vs Placebo; Test type: Superiority; ANCOVA; Least squares means = -38.7, 95% CI 2-sided [-54.29 to -23.11]

3. Secondary Outcome: Total Pain Relief (TOTPAR)
Description: Pain relief was measured using Categorical Pain Relief Rating Scale (0 = No relief, 1 = a little relief, 2 = some relief, 3 = a lot of relief, 4 = complete relief). Total pain relief scores (TOTPARs) were calculated by multiplying the pain relief score at each postdose time point by the duration (in hours) since the preceding time point and then summing these values.
Time Frame: Up to 24 hours
Population: Per-protocol population
Measure: Mean (Standard Deviation); unit: Scores on a scale * hours
Arm/Group | Naproxen Sodium (Aleve, BAY117031) | Ibuprofen (Advil) | Placebo
Number analyzed (Participants) | 166 | 165 | 54
Scores on a scale * hours | 47.16 (28.228) | 28.96 (21.097) | 13.40 (23.328)
Statistical Analysis 1: Comparison: Naproxen Sodium (Aleve, BAY117031) vs Ibuprofen (Advil); Test type: Superiority; ANCOVA; Least squares means = -18.21, 95% CI 2-sided [-23.52 to -12.89]
Statistical Analysis 2: Comparison: Naproxen Sodium (Aleve, BAY117031) vs Placebo; Test type: Superiority; ANCOVA; Least squares means = -33.72, 95% CI 2-sided [-41.29 to -26.14]
Statistical Analysis 3: Comparison: Ibuprofen (Advil) vs Placebo; Test type: Superiority; ANCOVA; Least squares means = -15.51, 95% CI 2-sided [-23.09 to -7.93]

ADVERSE EVENTS:
Time Frame: From start of study drug up to 10 days after the administration of study drug
Groups:
- Naproxen Sodium (Aleve, BAY117031): Subjects received one single dose of 440 mg naproxen sodium tablets (200 mg x 2 tablets, oral) after randomization
- Placebo: Subjects received one single dose of matching placebo tablets (2 tablets, oral) after randomization
- Ibuprofen (Advil): Subjects received one single dose of 400 mg ibuprofen tablets (200 mg x 2 tablets, oral) after randomization
Arm/Group | Naproxen Sodium (Aleve, BAY117031) | Placebo | Ibuprofen (Advil)
All-Cause Mortality (participants affected / at risk) | 0/166 | 0/55 | 0/166
Serious Adverse Events (participants affected / at risk) | 1/166 | 0/55 | 0/166
Other Adverse Events (participants affected / at risk) | 25/166 | 16/55 | 31/166
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Naproxen Sodium (Aleve, BAY117031) (N=166) | Placebo (N=55) | Ibuprofen (Advil) (N=166)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Naproxen Sodium (Aleve, BAY117031) (N=166) | Placebo (N=55) | Ibuprofen (Advil) (N=166)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Eye pain (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Eye swelling (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Aphthous ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Breath odour (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 9 (10) | 11 (12) | 17 (20)
Paraesthesia oral (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 7 (10) | 7 (9)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 1 (1)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Alveolar osteitis (Infections and infestations) | 4 (4) | 0 (0) | 1 (1)
Ear infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Periodontitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Incision site pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 4 (5) | 1 (1) | 5 (5)
Headache (Nervous system disorders) | 3 (3) | 7 (7) | 6 (6)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Nervousness (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-02-15): https://cdn.clinicaltrials.gov/large-docs/06/NCT03404206/Prot_000.pdf
  • Statistical Analysis Plan (2018-08-24): https://cdn.clinicaltrials.gov/large-docs/06/NCT03404206/SAP_001.pdf